CLINICAL TRIAL: NCT00755365
Title: Intraoperative Angioembolization in the Management of Pelvic Fracture-Related Hemodynamic Instability
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, J. Spence Reid, Principal Investigator, Milton S. Hershey Medical Center
Other Study IDs: 28576EM
Record Dates: First submitted 2008-09-16; First posted 2008-09-18 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Pelvic Fractures and Associated Hemodynamic Instability
Keywords: pelvic fractures; angioembolism; Treatment at Hershey Medical Center; Angioembolization in Operating Room
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Mortality associated with pelvic fractures resulting from blunt trauma ranges between 6 and 18%. In cases where hemodynamic instability is also present, the mortality rate is significantly greater, and has been reported as high as 60%. There is no general consensus among traumatologists as to the initial management of this complicated subgroup of patients. It is largely debated whether emergent orthopedic fixation or angiographic embolization should be the first line of treatment for pelvic hemorrhage

DETAILED DESCRIPTION:
Pelvic fractures are not usually isolated injuries and it is common that these severely injured patients have concomitant abdominal or thoracic trauma further complicating their management. In situations where multiple sources of hemodynamic instability exist, the need to control hemorrhage quickly becomes imperative. In patients where emergent laparotomy or thoracotomy is indicated, the time until pelvic bleeding sources are addressed is prolonged. Some would argue that the best initial management of the pelvic fractures should be surgical stabilization, while others would support immediate angioembolization of actively bleeding pelvic vessels. The main drawback of angiographic embolization is that it occurs in a separate Angio Suite facility, with concerns being time lost to patient transport and an environment less capable of managing these extremely unstable patients.

At Hershey Medical Center, ten patients suffering pelvic fractures with associated hemodynamic instability between 2003 and 2007 were managed with intraoperative angioembolization (in the Operating Room as opposed to the Angio Suite). Extensive review of published orthopaedic, trauma surgery, and radiology journals yielded no other literature regarding intraoperative angioembolization as a management approach for these patients. Whether or not this approach has been carried out at other medical institutions, it is undoubtedly rare and results have yet to be reported in widely available literature. This novel approach has the potential to stop pelvic bleeding sooner and in a more controlled environment, where surgical stabilization can also be accomplished simultaneously. Statistical analysis and review of these patients has not been done, but may possibly show improvements in survival, shorter length of hospital stay, less time to embolization, and decreased need for supportive measures such as blood or platelet transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pelvic fractures and associated hemodynamic instability
* Treatment at Hershey Medical Center
* Patient management involved angioembolization in Operating Room

Exclusion Criteria:

* Patients below 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects in this study are trauma patients over 18 years of age who suffered pelvic fractures and developed associated hemodynamic instability between January 1, 2003 and December 31, 2007. All patients were treated at Hershey Medical Center and received intraoperative angioembolization as a part of their medical management.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
To present intraoperative angioembolization as a option in management of this group of patients and to describe the outcomes of these ten patients | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Soence Reid, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Agolini SF, Shah K, Jaffe J, Newcomb J, Rhodes M, Reed JF 3rd. Arterial embolization is a rapid and effective technique for controlling pelvic fracture hemorrhage. J Trauma. 1997 Sep;43(3):395-9. doi: 10.1097/00005373-199709000-00001. PMID 9314298
- [Background] Balogh Z, King KL, Mackay P, McDougall D, Mackenzie S, Evans JA, Lyons T, Deane SA. The epidemiology of pelvic ring fractures: a population-based study. J Trauma. 2007 Nov;63(5):1066-73; discussion 1072-3. doi: 10.1097/TA.0b013e3181589fa4. PMID 17993952
- [Background] Balogh Z, Caldwell E, Heetveld M, D'Amours S, Schlaphoff G, Harris I, Sugrue M. Institutional practice guidelines on management of pelvic fracture-related hemodynamic instability: do they make a difference? J Trauma. 2005 Apr;58(4):778-82. doi: 10.1097/01.ta.0000158251.40760.b2. PMID 15824655
- [Background] Bassam D, Cephas GA, Ferguson KA, Beard LN, Young JS. A protocol for the initial management of unstable pelvic fractures. Am Surg. 1998 Sep;64(9):862-7. PMID 9731815
- [Background] Fangio P, Asehnoune K, Edouard A, Smail N, Benhamou D. Early embolization and vasopressor administration for management of life-threatening hemorrhage from pelvic fracture. J Trauma. 2005 May;58(5):978-84; discussion 984. doi: 10.1097/01.ta.0000163435.39881.26. PMID 15920412
- [Background] Miller PR, Moore PS, Mansell E, Meredith JW, Chang MC. External fixation or arteriogram in bleeding pelvic fracture: initial therapy guided by markers of arterial hemorrhage. J Trauma. 2003 Mar;54(3):437-43. doi: 10.1097/01.TA.0000053397.33827.DD. PMID 12634521
- [Background] Sadri H, Nguyen-Tang T, Stern R, Hoffmeyer P, Peter R. Control of severe hemorrhage using C-clamp and arterial embolization in hemodynamically unstable patients with pelvic ring disruption. Arch Orthop Trauma Surg. 2005 Sep;125(7):443-7. doi: 10.1007/s00402-005-0821-7. PMID 15977021